CLINICAL TRIAL: NCT00912847
Title: Validity and Cost-Effectiveness of a New Screening Test for Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Prof. Tony Mok, Clinical Oncology
Other Study IDs: RHCC002
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2009-06-03 (Estimated); Status verified 2009-06

CONDITIONS: Hepatitis B Virus
Keywords: HBV carriers
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- JHC: AFP > 20 ng/ml and USG positive
- Non JHC: patient without AFP > 20 or USG negative

SUMMARY:
The purpose of this study is:

1. To establish and compare the diagnostic utilities for hepatocellular carcinoma (HCC) screening tests of (a) HS-AFP, (b) AFP + US,(c) AFP alone and (d) US alone (within HBV carriers between age 40 and 70 years);
2. To establish the cost-effectiveness of the screening tests;
3. To compare tumor sizes, resection rates, and survival rates up to 18 months between those who were screened by HS-AFP those of a historical control group that was not screened.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 70 years
* Seropositive for HBsAg
* Child's A or B
* Life expectancy of more than 2 years

Exclusion Criteria:

* Non-HBV related cirrhosis
* History of malignancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HBV carriers between age 40 and 70 years
Sampling Method: Non-Probability Sample
Enrollment: 1018 (Actual)
Dates: Start 1997-10; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)